CLINICAL TRIAL: NCT03089723
Title: Comparative Study of the Intraarticular Treatment of Carpometacarpal Joint Ostearthritis of the Thumb With Lavage With Saline Solution, or Lavage and Injection of Hyaluronic Acid and Mannitol.
Brief Title: Saline Lavage X Saline Lavage and Osteonil® Mini in Rizarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, MD; PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14733/16
Record Dates: First submitted 2017-01-12; First posted 2017-03-24 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Rhizarthrosis; Metabolic Disease
Keywords: carpometacarpal joint ostearthritis; hyaluronic acid; Rhizarthrosis
MeSH Terms: conditions — Metabolic Diseases | interventions — Range of Motion, Articular; Therapeutic Irrigation; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavage with Saline (LS) (Experimental): Under sterile conditions, the 1st carpometacarpal (CMC) will be locally anesthetized with ropivacaine and will be submitted to joint lavage with physiologic saline solution 2 to 5 mL (injection with a 30x8 needle and drained with the same needle after removal of the syringe. After emptying of the joint, 1mL saline solution will be injected.
  Patients will ask to answer Visual Analog Scale (VAS) questionnaire, Range of Motion (ROM), Quick DASH, Sollerman Test, and functional grip strength (palmar grip strength, lateral grip strength and pulp-pulp pinch strength) evaluations immediately prior to the procedure and after 1, 3 and 6 months of each joint.
  Interventions: Behavioral: Visual Analog Scale (VAS); Behavioral: Range of Motion (ROM); Behavioral: Palmar grip strength; Behavioral: Lateral grip strength; Behavioral: Pulp-pulp pinch strength; Drug: Lavage with physiologic saline solution; Behavioral: Quick Dash; Behavioral: Sollerman Test
- Lavage with Osteonil® Mini (LO) (Experimental): Under sterile conditions, the 1st carpometacarpal (CMC) will be locally anesthetized with ropivacaine and will be submitted to lavage with physiologic saline solution and Osteonil® Mini 1mL of 10mg will be injected in the 1st CMC joint.
  Patients will ask to answer Visual Analog Scale (VAS) questionnaire, Range of Motion (ROM), Quick DASH, Sollerman Test, and functional grip strength (palmar grip strength, lateral grip strength and pulp-pulp pinch strength) evaluations immediately prior to the procedure and after 1, 3 and 6 months of each joint.
  Interventions: Behavioral: Visual Analog Scale (VAS); Behavioral: Range of Motion (ROM); Behavioral: Palmar grip strength; Behavioral: Lateral grip strength; Behavioral: Pulp-pulp pinch strength; Drug: Lavage with physiologic saline solution and Osteonil® Mini; Behavioral: Quick Dash; Behavioral: Sollerman Test

INTERVENTIONS:
Behavioral: Visual Analog Scale (VAS) — Answer Visual Analog Scale (VAS) questionnaire at baseline, 1 month, 3 months and 6 months
Behavioral: Range of Motion (ROM) — submitted to ROM at at baseline, 1 month, 3 months and 6 months
Behavioral: Palmar grip strength — submitted to palmar grip strength at at baseline, 1 month, 3 months and 6 months
Behavioral: Lateral grip strength — submitted to lateral grip strength at at baseline, 1 month, 3 months and 6 months
Behavioral: Pulp-pulp pinch strength — submitted to pulp-pulp pinch strength strength at at baseline, 1 month, 3 months and 6 months
Drug: Lavage with physiologic saline solution — Joint lavage with physiologic saline solution. After emptying of the joint, 1mL saline solution will be injected.
  Other Names: Lavage with Saline (LS)
  Arms: Lavage with Saline (LS)
Drug: Lavage with physiologic saline solution and Osteonil® Mini — Joint lavage with physiologic saline solution and Osteonil® Mini
  Other Names: Lavage with Osteonil® Mini (LO)
  Arms: Lavage with Osteonil® Mini (LO)
Behavioral: Quick Dash — Answer Quick Dash questionnaire at baseline, 1 month, 3 months and 6 months
Behavioral: Sollerman Test — Perform Sollerman Test at baseline, 1 month, 3 months and 6 months

SUMMARY:
Although a common problem, hand osteoarthritis (HOA) is less studied than knee and hip. In the age group of 71-100 years, the prevalence of symptomatic HOA reaches 26% of women and 13% of men. These patients lose hand strength and have difficulty with day-to-day manual activities. The main joints involved are the proximal and distal interphalangeals and the carpometacarpal joint of the thumb. In the educational Project PARQVE, the prevalence of HOA was 23.7% at inclusion in the program, and 47.4% after one year, with loss of grip strength. There is controversy over the effect of viscosupplementation in the treatment of rhizarthritis when considering pain. However, strength is a very important function parameter that must be evaluated for function and quality of life maintenance. Concerned about the importance of maintaining strength and function in our program (PARQVE), we have added specific exercises tom improve hand strength and range of motion. Trying to optimize the treatment and confronting questions about the effect of the joint wash, called placebo in the comparative studies with corticosteroid and/or hyaluronic acid injection, we did a work where all the patients will be washed with physiological saline solution but a group, after emptying, will receive 1mL of hyaluronic acid with mannitol.

PURPOSE: To compare isolated lavage with lavage followed by injection of hyaluronic acid with mannitol into carpometacarpal osteoarthritis joint of the thumb.

METHODS: Forty joints of patients with multiple osteoarthritis (rhizoarthritis, including) and comorbidities (two or more of: overweight or obesity, hyperglycemia, dyslipidemia, hyperuricemia, hypertension) will be allocated into two groups: Lavage (LS) and Lavage and Injection Hilauronic acid (LO). Both groups will undergo joint lavage with saline solution. The LO group will receive the 20 mg / mL hilauronic acid injection with 5mg mannitol. Both groups will be guided in the clinical treatment of osteoarthritis and metabolic syndrome and will be given daily exercises for the hands. They will be evaluated with the quick DASH questionnaire, Sollerman Test and by measuring the palmar, lateral and pulp-pulp grip strength, in addition to measuring the ROM and VAS pain moments immediately prior to the procedure, one, three and six months after the articular procedure.

DETAILED DESCRIPTION:
Patients with multiple osteoarthritis (including carpometacarpal joint of the thumb, stages I to III - Eaton et al.) in treatment at the Institute of Orthopedics and Traumatology fo the Clinics Hospital - University of São Paulo (IOT-HC-FMUSP) will be invited to participate in this study.

All patients are obliged to participate in a two-day education course on OA. During the program they are instructed about OA, metabolic syndrome, comorbidities and importance of diet, and daily exercise (including specific exercises for the hand).

After inclusion, 40 joints will be randomized in one of two treatment options, i.e., Lavage with saline solution and final injection of 1mL of saline solution, or lavage with saline solution followed by injection of 10mg of hyaluronic acid with mannitol (5mg).

After the procedure patients will receive naproxen 500mg twice daily for 5 days.

Patients will be instructed to exercise at least 180 minutes/week and if possible daily exercise for the hand (5 to 10 minutes daily).

Patients will be instructed to write down when and what they exercised as well as their daily medication intake (for co-morbidities and pain).

All patients will be submitted to pain (VAS), range of motion (ROM), Quick DASH, Sollermand Test and functional (palmar grip strength and lateral and pulp-pulp pinch strength) evaluations immediately prior to the procedure and after 1, 3 and 6 months of each joint.

As the assessments of pain, range of motion and strength will be compared with measurements of the same limb at inclusion, each hand involved of the patient will be considered as a case.

The "n" was calculated to obtain a statistical power of 80% and a level of significance of 5%. To do this, we considered the mean and standard deviation of the pulp-pulp pinch (our primary outcome) found in previous study of the prevalence of hand OA in individuals with knee osteoarthritis submitted to our educational program. A sample size was used to detect a variation of 1 point on the two-tailed pulp-pulp pinches. The sample size calculated by group was 16. Considering also possible faults and abandon of about 20% of the patients, the value of 20 patients per group was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with multiple arthritis (including CMC OA of the thumb) with comorbidities (metabolic syndrome, i.e., OA and overweight / obesity, and/or hyperglycemia, and/or dyslipidemia, and/or hyperuricemia, and/or hypertension).
* CMC OA joint of the thumb stages I to III as classified by Eaton et al. (4)

Exclusion Criteria:

* Missing classes or functional evaluations
* Not performing the exercises as instructed

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in grip strength at 6 months | Baseline, 1 month, 3 months and 6 months.
  Perform test and collected data in baseline, 1 month, 3 months and 6 months.

SECONDARY OUTCOMES:
Assess improvement in pain | Baseline, 1 month, 3 months and 6 months.
  Answer VAS (Visual Analog Scale)
Assess improvement in range of motion | Baseline, 1 month, 3 months and 6 months.
  Measure range of motion
Assess improvement in palmar grip strength | Baseline, 1 month, 3 months and 6 months.
  Perform palmar grip strength
Assess improvement in lateral pinch strength. | Baseline, 1 month, 3 months and 6 months.
  Perform lateral pinch strength.
Assess improvement in Pulp-pulp pinch strength | Baseline, 1 month, 3 months and 6 months.
  Perform pulp-pulp pinch strength

CONTACTS AND LOCATIONS:
Overall Officials: Marcia U Rezende, MD; PhD, Principal Investigator — Department of Orthopedics and Traumatology - HCFMUSP
Locations (1):
- Instituto de Ortopedia e Traumatologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kennedy CD, Manske MC, Huang JI. Classifications in Brief: The Eaton-Littler Classification of Thumb Carpometacarpal Joint Arthrosis. Clin Orthop Relat Res. 2016 Dec;474(12):2729-2733. doi: 10.1007/s11999-016-4864-6. Epub 2016 May 4. No abstract available. PMID 27146653
- [Background] Gillis J, Calder K, Williams J. Review of thumb carpometacarpal arthritis classification, treatment and outcomes. Can J Plast Surg. 2011 Winter;19(4):134-8. doi: 10.1177/229255031101900409. PMID 23204884
- [Background] Gehrmann SV, Tang J, Li ZM, Goitz RJ, Windolf J, Kaufmann RA. Motion deficit of the thumb in CMC joint arthritis. J Hand Surg Am. 2010 Sep;35(9):1449-53. doi: 10.1016/j.jhsa.2010.05.026. PMID 20807622
- [Background] Eaton RG, Lane LB, Littler JW, Keyser JJ. Ligament reconstruction for the painful thumb carpometacarpal joint: a long-term assessment. J Hand Surg Am. 1984 Sep;9(5):692-99. doi: 10.1016/s0363-5023(84)80015-5. PMID 6491213
- [Background] Matullo KS, Ilyas A, Thoder JJ. CMC arthroplasty of the thumb: a review. Hand (N Y). 2007 Dec;2(4):232-9. doi: 10.1007/s11552-007-9068-9. Epub 2007 Aug 7. PMID 18780059
- [Background] Diaconu M, Mathoulin C, Facca S, Liverneaux P. Arthroscopic interposition arthroplasty of the trapeziometacarpal joint. Chir Main. 2011 Sep;30(4):282-7. doi: 10.1016/j.main.2011.06.009. Epub 2011 Jul 19. PMID 21816649
- [Background] Vermeulen GM, Slijper H, Feitz R, Hovius SE, Moojen TM, Selles RW. Surgical management of primary thumb carpometacarpal osteoarthritis: a systematic review. J Hand Surg Am. 2011 Jan;36(1):157-69. doi: 10.1016/j.jhsa.2010.10.028. PMID 21193136
- [Background] Bell R, Desai S, House H, O'Donovan T, Palmer AK. A retrospective multicenter study of the Artelon(R) carpometacarpal joint implant. Hand (N Y). 2011 Dec;6(4):364-72. doi: 10.1007/s11552-011-9366-0. Epub 2011 Sep 24. PMID 23204961
- [Background] Badia A, Sambandam SN. Total joint arthroplasty in the treatment of advanced stages of thumb carpometacarpal joint osteoarthritis. J Hand Surg Am. 2006 Dec;31(10):1605-14. doi: 10.1016/j.jhsa.2006.08.008. PMID 17145380
- [Background] Sillem H, Backman CL, Miller WC, Li LC. Comparison of two carpometacarpal stabilizing splints for individuals with thumb osteoarthritis. J Hand Ther. 2011 Jul-Sep;24(3):216-25; quiz 126; discussion 227-30. doi: 10.1016/j.jht.2010.12.004. Epub 2011 Mar 21. PMID 21420278
- [Background] Valdes K, von der Heyde R. An exercise program for carpometacarpal osteoarthritis based on biomechanical principles. J Hand Ther. 2012 Jul-Sep;25(3):251-62; quiz 263. doi: 10.1016/j.jht.2012.03.008. PMID 22794499
- [Background] Clegg TE, Caborn D, Mauffrey C. Viscosupplementation with hyaluronic acid in the treatment for cartilage lesions: a review of current evidence and future directions. Eur J Orthop Surg Traumatol. 2013 Feb;23(2):119-24. doi: 10.1007/s00590-012-0940-0. Epub 2012 Jan 28. PMID 23412441
- [Background] Gigante A, Callegari L. The role of intra-articular hyaluronan (Sinovial) in the treatment of osteoarthritis. Rheumatol Int. 2011 Apr;31(4):427-44. doi: 10.1007/s00296-010-1660-6. Epub 2010 Nov 28. PMID 21113807
- [Background] Fakhari A, Berkland C. Applications and emerging trends of hyaluronic acid in tissue engineering, as a dermal filler and in osteoarthritis treatment. Acta Biomater. 2013 Jul;9(7):7081-92. doi: 10.1016/j.actbio.2013.03.005. Epub 2013 Mar 15. PMID 23507088
- [Background] Mei-Dan O, Carmont M, Laver L, Mann G, Maffulli N, Nyska M. Intra-articular injections of hyaluronic acid in osteoarthritis of the subtalar joint: a pilot study. J Foot Ankle Surg. 2013 Mar-Apr;52(2):172-6. doi: 10.1053/j.jfas.2012.12.008. Epub 2013 Jan 17. PMID 23333279
- [Background] de Campos GC, Rezende MU, Pailo AF, Frucchi R, Camargo OP. Adding triamcinolone improves viscosupplementation: a randomized clinical trial. Clin Orthop Relat Res. 2013 Feb;471(2):613-20. doi: 10.1007/s11999-012-2659-y. Epub 2012 Oct 26. PMID 23100188
- [Background] Heyworth BE, Lee JH, Kim PD, Lipton CB, Strauch RJ, Rosenwasser MP. Hylan versus corticosteroid versus placebo for treatment of basal joint arthritis: a prospective, randomized, double-blinded clinical trial. J Hand Surg Am. 2008 Jan;33(1):40-8. doi: 10.1016/j.jhsa.2007.10.009. PMID 18261664
- [Background] Frizziero A, Maffulli N, Masiero S, Frizziero L. Six-months pain relief and functional recovery after intra-articular injections with hyaluronic acid (mw 500-730 KDa) in trapeziometacarpal osteoarthritis. Muscles Ligaments Tendons J. 2014 Jul 14;4(2):256-61. eCollection 2014 Apr. PMID 25332944
- [Background] Bahadir C, Onal B, Dayan VY, Gurer N. Comparison of therapeutic effects of sodium hyaluronate and corticosteroid injections on trapeziometacarpal joint osteoarthritis. Clin Rheumatol. 2009 May;28(5):529-33. doi: 10.1007/s10067-008-1079-6. Epub 2009 Jan 10. PMID 19137353
- [Background] Kroon FP, Rubio R, Schoones JW, Kloppenburg M. Intra-Articular Therapies in the Treatment of Hand Osteoarthritis: A Systematic Literature Review. Drugs Aging. 2016 Feb;33(2):119-33. doi: 10.1007/s40266-015-0330-5. PMID 26650235
- [Background] Campos GC, Kohara MT, Rezende MU, Santana OF, Moreira MM, Camargo OP. Schooling of the patients and clinical application of questionnaires in osteoarthitis. Acta Ortop Bras. 2014;22(5):256-9. doi: 10.1590/1413-78522014220500980. PMID 25328433
- [Background] de Rezende MU, Hissadomi MI, de Campos GC, Frucchi R, Pailo AF, Pasqualin T, Brito NL, Santana OF, Moreira MM, Strutz CG, Matos NB, de Camargo OP, Hernandez AJ. One-Year Results of an Educational Program on Osteoarthritis: A Prospective Randomized Controlled Trial in Brazil. Geriatr Orthop Surg Rehabil. 2016 Jun;7(2):86-94. doi: 10.1177/2151458516645634. Epub 2016 May 11. PMID 27239382
- [Background] Mendoza G, Alvarez AI, Pulido MM, Molina AJ, Merino G, Real R, Fernandes P, Prieto JG. Inhibitory effects of different antioxidants on hyaluronan depolymerization. Carbohydr Res. 2007 Jan 15;342(1):96-102. doi: 10.1016/j.carres.2006.10.027. Epub 2006 Nov 2. PMID 17123492
- [Background] Vad VB, Bhat AL, Sculco TP, Wickiewicz TL. Management of knee osteoarthritis: knee lavage combined with hylan versus hylan alone. Arch Phys Med Rehabil. 2003 May;84(5):634-7. doi: 10.1016/s0003-9993(02)04811-6. PMID 12736873